CLINICAL TRIAL: NCT06745999
Title: A Single Center, Observational Study to Evaluate the Effectiveness and Safety of Cryotherapy in Combination with 10% ALA Gel Red Light PDT in the Treatment of Actinic Keratosis on the Full Face.
Brief Title: Cryotherapy in Combination with Red Light PDT for Actinic Keratosis of Full Face
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Psoriasis Treatment Center of Central New Jersey (Other)
Collaborators: Biofrontera Bioscience GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PTC11
Record Dates: First submitted 2024-12-18; First posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-03

CONDITIONS: Actinic Keratoses
MeSH Terms: conditions — Keratosis, Actinic | interventions — Aminolevulinic Acid; Gels; Photochemotherapy; Cryotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- cryotherapy followed by 10% ALA gel Red light PDT (Experimental)
  Interventions: Drug: Ameluz 10% Topical Gel; Device: Red Light PDT; Procedure: Cryotherapy
- 10% ALA gel Red Light PDT followed by cryotherapy (Experimental)
  Interventions: Drug: Ameluz 10% Topical Gel; Device: Red Light PDT; Procedure: Cryotherapy

INTERVENTIONS:
Drug: Ameluz 10% Topical Gel — Paired with device intervention of red light PDT
  Other Names: ALA gel
Device: Red Light PDT — Paired with drug intervention of Ameluz 10% topical gel
Procedure: Cryotherapy — Liquid Nitrogen

SUMMARY:
40 patients randomized 1:1 to receive cryotherapy followed by 10% ALA gel Red light PDT vs. to 10% ALA gel Red Light PDT followed by cryotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adult ≥ 18 years of age;
2. 6-12 actinic keratosis grade I, II, and III on the full face.
3. Willing to avoid excessive sunlight or ultraviolet (UV) light exposure, including the use of tanning beds, to the face or scalp during study participation.
4. Females of childbearing potential (FCBP) must have a negative serum pregnancy test at Screening and negative urine pregnancy test at Baseline. FCBP who engage in activity in which conception is possible must use one of the approved contraceptive options: hormonal contraception; intrauterine device (IUD); tubal ligation; or partner's vasectomy; Male or female condom diaphragm with spermicide, cervical cap with spermicide, or contraceptive sponge with spermicide.
5. Able and willing to give written informed consent prior to performance of any study-related procedures

Exclusion Criteria:

1. Presence of other skin conditions that may affect the study participant, investigator's ability to assess treatment, or intolerance to any ingredient in 10% ALA gel.
2. Treatment with 5-fluorouracil (5-FU), imiquimod, ingenol mebutate, diclofenac, photodynamic therapy, or other topicals and treatments for AK within the treatment area or within 2 cm of the treatment area, within 12 weeks of baseline.
3. Use of liquid nitrogen, excision, curettage, dermabrasion, chemical peel or laser resurfacing in the treatment area within 60 days.
4. Use of systemic retinoids (eg, isotretinoin, acitretin) within 6 months
5. Women of childbearing potential who are pregnant, intend to become pregnant, or are lactating.
6. Use of any investigational drug within 4 weeks prior to enrollment or within 5 pharmacokinetic/pharmacodynamic half-lives, if known (whichever is longer).
7. Any clinically significant (as determined by the Investigator) cardiac, endocrinologic, pulmonary, neurologic, psychiatric, hepatic, renal, hematologic, immunologic disease, or other major disease that is currently uncontrolled.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-05-03 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Percentage change in total lesions at Week 24 | 24 Weeks
  Percentage change From Baseline in Total Lesion Complete Response at Week 24

CONTACTS AND LOCATIONS:
Locations (1):
- Psoriasis Treatment Center of New Jersey, East Windsor, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided